CLINICAL TRIAL: NCT06561906
Title: Establish Diagnostic and Prognostic Models for Preclinical AD Patients Based on Multimodal MRI, Behavioral, Genetic, and Plasma Biomarkers
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-341-01
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease, Late Onset; Mild Cognitive Impairment; Subjective Cognitive Decline
Keywords: magnetic resonance imaging; spatial navigation; olfaction; genetic; plasma biomarkers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Spatial Navigation; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal control: Subjects without memory complaints and associated worries and do not meet the diagnostic criteria for mild cognitive impairment (MCI) are recruited as normal control (NC).
  Interventions: Other: Multimodal magnetic resonance imaging scanning, behavioral, genetic and plasma biomarker testing
- Subjective cognitive decline: Subjects who complain of memory decline within the last 5 years and express worries associated with memory decline and do not meet the diagnostic criteria for MCI are defined as subjective cognitive decline (SCD).
  Interventions: Other: Multimodal magnetic resonance imaging scanning, behavioral, genetic and plasma biomarker testing
- Mild cognitive impairment: Participants are considered MCI patients with scores >1 standard deviation (SD) below the normative means in both subtests within one cognitive domain or >1 SD below the normative means in three single tests in three different domains.
  Interventions: Other: Multimodal magnetic resonance imaging scanning, behavioral, genetic and plasma biomarker testing
- Alzheimer's disease dementia: Patients are diagnosed as AD dementia by an experienced neurologist based on MMSE and CSF/PET biomarker evidence.
  Interventions: Other: Multimodal magnetic resonance imaging scanning, behavioral, genetic and plasma biomarker testing

INTERVENTIONS:
Other: Multimodal magnetic resonance imaging scanning, behavioral, genetic and plasma biomarker testing — Multimodal magnetic resonance imaging scanning, including 3DT1, 3DT2, 3DFLAIR, functional MRI, DTI, NODDI, ASL, QSM behavioral testing, such as olfaction and spatial navigation genetic testing, such as APOE, BDNF plasma biomarker testing, such as ptau, Aβ42/40、NfL、GFAP

SUMMARY:
To establish the diagnostic and prognostic models that could help the preclinical identification of subjects at higher risk of clinical progression to mild cognitive impairment and dementia based on combined features of baseline demographic, cognitive, behavioral, multimodal MRI, genetic, and plasma data.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a global concern. Due to the lack of effective therapeutic methods targeting late-stage AD patients, it is critical to investigate brain alterations in the preclinical stage to pave the way for early diagnosis and intervention. Structural and functional magnetic resonance imaging (MRI) has been proven to be an effective and non-invasive approach to explore the neural mechanisms underlying neurological disorders. Genetic factors such as apolipoprotein E and plasma biomarkers play important roles in AD development and progression. However, the interaction effects of risk genes and different pathologic pathways implicated in the pathogenesis of AD remain unclear. Furthermore, the diagnostic and prognostic models that could predict future cognitive decline or clinical progression based on objective features derived from baseline demographic, cognitive, behavioral, multimodal MRI, genetic, and plasma data need to be further explored.

We aim to investigate the neural basis underlying early cognitive deficits using structural and functional MRI data combined with novel analytical methods such as dynamic functional connectivity, surface-based morphometry, graph theory, multilayer network, functional-structural coupling, hidden Markov model, and connectome gradient mapping. Secondly, to explore the interaction effects of risk genes, which may help a better illustration of different biological pathways implicated in the pathogenesis of Alzheimer's disease. Thirdly, to investigate the divergent and dynamic abnormalities of multimodal imaging markers across different stages of Alzheimer's disease and their associations with plasma biomarkers, which may enhance our understanding of the neuropathological mechanisms. Fourthly, to provide scientific evidence on the potential targets for early intervention of neurodegenerative diseases. Lastly, to establish the diagnostic and prognostic models that could help the preclinical identification of subjects at higher risk of clinical progression to mild cognitive impairment and dementia based on combined features of baseline multimodal biomarkers. These studies may help a better understanding of the neural and biological basis underlying AD and pave the way for early diagnosis and intervention.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were 50-79 years old and having 8 or more years of education.

Exclusion Criteria:

* Participants with a history of stroke, other neurological disorders that could lead to cognitive impairment (Parkinson's disease, encephalitis, epilepsy, brain tumors, etc.), severe anxiety or depression, and contraindications for magnetic resonance imaging (MRI) were not enrolled.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese Han nationality
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the area under the curve of the classification analysis between progressors and nonprogressors | Baseline, Year 1, Year 2, Year 3
  We'll measure the area under the curve of the ROC curves based on combined features of baseline demographic, cognitive, behavioral, multimodal MRI, genetic, and plasma data in discriminating those convert to MCI or AD (progressors) from those do not convert (nonprogressors)

SECONDARY OUTCOMES:
mediation effects of MRI on the associations between gene/plasma biomarker and cognition/behavior | Baseline
  We'll explore whether MRI features could act as mediators between genetic factors and cognition or behavior, as well as between plasma biomarkers and cognition or behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to the clinical nature of the data, the data that support the findings of this study are not freely available but can be made available by the corresponding author, upon reasonable request. A formal data-sharing agreement is needed before any data can be shared.

REFERENCES:
- [Background] Chen Q, Chen F, Long C, Zhu Y, Jiang Y, Zhu Z, Lu J, Zhang X, Nedelska Z, Hort J, Zhang B. Spatial navigation is associated with subcortical alterations and progression risk in subjective cognitive decline. Alzheimers Res Ther. 2023 Apr 25;15(1):86. doi: 10.1186/s13195-023-01233-6. PMID 37098612